CLINICAL TRIAL: NCT02379923
Title: The Asahi Intecc PTCA Chronic Total Occlusion Study
Acronym: CTO-PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asahi Intecc USA Inc (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIUCT-001
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease; Coronary Artery Chronic Total Occlusion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Crossing of Coronary Artery CTO (Experimental): This is a single arm intent to treat study. A subject is considered enrolled when the subject has given informed consent and meets all inclusion and exclusion criteria, including angiographic inclusion and exclusion criteria, which includes an attempt to cross the target lesion with an investigational device (ASAHI PTCA Guidewire or ASAHI Corsair Microcatheter). Clinical evaluation up to hospital discharge is conducted on all enrolled subjects. The purpose of the clinical follow-up is to determine if the subject has experienced or is experiencing any adverse events
  Interventions: Device: Crossing of Coronary Artery CTO

INTERVENTIONS:
Device: Crossing of Coronary Artery CTO — Standard angiographic procedures will be followed for this study. The primary objective of this trial is to evaluate confirmation of placement of any guidewire beyond the chronic total occlusion (CTO) in the true vessel lumen in patients in which at least one Asahi series of guidewires and/or Corsair microcatheter were used.
  Procedure success will be defined as angiographic visualization of any guidewire in a position either distal or proximal to the occlusion depending on the route of access and the absence of in-hospital MACE.
  Other Name: ASAHI Corsair Microcatheter, ASAHI PTCA Guide Wires
  Other Names: Corsair, Gaia, Asahi Guide Wires

SUMMARY:
The primary objective of this trial is to evaluate confirmation of placement of any guidewire beyond the chronic total occlusion (CTO) in the true vessel lumen in patients in which at least one Asahi series of guidewires and/or Corsair microcatheter were used.

Procedure success will be defined as angiographic visualization of any guidewire in a position either distal or proximal to the occlusion depending on the route of access and the absence of in-hospital major adverse cardiac events (MACE).

DETAILED DESCRIPTION:
This prospective, multi-center, single-arm, intent-to-treat (ITT) study is designed to assess the safety and effectiveness of the investigational products for the treatment of CTOs in a native coronary artery.

The primary objective of this trial is to evaluate confirmation of placement of any guidewire beyond the CTO in the true vessel lumen in patients in which at least one Asahi series of guidewires and/or Corsair microcatheter were used.

The population for this study is subjects with signs and/or symptoms considered typical of ischemic heart disease attributed to a CTO in a native coronary artery, who are suitable for a percutaneous revascularization.

Procedure success will be defined as angiographic visualization of any guidewire in a position either distal or proximal to the occlusion depending on the route of access and the absence of in-hospital major adverse cardiac events (MACE). All subjects are followed through hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria:

  1. Subject is ≥ 18 years of age at the time of consent
  2. Subject is experiencing clinical symptoms considered suggestive of ischemic heart disease (e.g., chest pain or discomfort, heart failure, etc.) or has evidence of myocardial ischemia (e.g., abnormal functional study) attributed to the CTO target vessel and is scheduled for clinically indicated percutaneous revascularization
  3. Subject is eligible and consents to undergo PCI procedure
  4. Subject is an acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA), stenting, and emergency coronary artery bypass grafting (CABG)
  5. Subject is willing and able to sign an Informed Consent Form approved by a local Institutional Review Board
  6. Female subjects of child-bearing potential must have a negative qualitative or quantitative pregnancy test within 7 days before the study procedure

     Angiographic Inclusion Criteria:
  7. A minimum of one de novo lesion with at least one target segment in a native coronary vessel meeting definition of chronic total occlusion. Non-study lesions will be treated first. A "chronic total occlusion" is any non-acute total coronary occlusion fulfilling the angiographic characteristics consistent with high-grade native coronary stenosis (TIMI 0) and estimated in duration at least 3 months by clinical history and/or comparison with antecedent angiogram or electrocardiogram. An attempt to cross the target lesion with at least one Asahi guidewire or a Corsair microcatheter must be made.

Exclusion Criteria:

* General Exclusion Criteria:

  1. Subjects with any history of allergy to iodinated contrast that cannot be effectively managed medically
  2. Evidence of acute Myocardial Infarction (MI) within 72 hours of the intended treatment defined as cardiac enzymes greater than Upper Limit of Normal (ULN).
  3. Previous coronary interventional procedure of any kind within the 30 days prior to the procedure
  4. Any contraindication to cardiac catheterization or to any of the standard concomitant therapies used during routine cardiac catheterization and PCI (e.g., aspirin, clopidogrel, unfractionated heparin, etc.)
  5. Target lesion requires treatment with a device after successful crossing other than PTCA prior to stent placement
  6. Subjects with known history of clinically significant abnormal laboratory findings including:

     * Neutropenia (<1000 neutrophils/mm3) within the previous 2 weeks
     * Thrombocytopenia (<100,000 platelets/mm3)
     * AST, ALT, alkaline phosphatase, or bilirubin > 1.5 × ULN
     * Serum creatinine > 2.0 mg/dL
  7. Subjects with evidence of ongoing or active clinical instability including the following:

     * Sustained systolic blood pressure < 100 mmHg or cardiogenic shock
     * Acute pulmonary edema or severe congestive heart failure
     * Suspected acute myocarditis, pericarditis, endocarditis, or cardiac tamponade
     * Suspected dissecting aortic aneurysm
     * Hemodynamically significant valvular heart disease, hypertrophic cardiomyopathy, restrictive cardiomyopathy, or congenital heart disease
  8. History of stroke or transient ischemic attack within the prior 6 months
  9. Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months
  10. History of bleeding diathesis or coagulopathy or refusal of blood transfusions
  11. Subjects with any other pathology such as cancer, mental illness, etc., which in the opinion of the Investigator, might put the patient at risk, preclude follow-up, or in any way confound the results of the study
  12. Known previous medical condition yielding expected survival less than 1 year
  13. Subjects who are unable or unwilling to comply with the protocol or not expected to complete the study period, including its follow-up requirements
  14. Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints;

      Angiographic Exclusion Criteria:
  15. Occlusion involves segment within previous stent
  16. Extensive lesion-related thrombus (TIMI thrombus grade 3 or 4)
  17. Previous stenting (drug-eluting or bare metal) in the target vessel unless the following conditions are met:

      * It has been at least 9 months since the previous stenting
      * That target lesion is at least 15 mm away from the previously placed stent
      * The previously stented segment (stent plus 5 mm on either side) has no more than 40% diameter stenosis, based on visual estimate
  18. The target vessel has other lesions proximal to the total occlusion identified with greater than 75% diameter stenosis based on visual estimate. However, planned stenting of the lesion in target vessel which is proximal to the target lesion and can be covered by a single stent (i.e., tandem lesions) are acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Heart Institute; Aaron Grantham, MD, Principal Investigator — MidAmerica Heart Institute
Locations (12):
- United States (12):
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Medical Center of the Rockies, Loveland, Colorado
  - Piedmont Healthcare, Atlanta, Georgia
  - Advocate Health and Hospitals Corp., Oakbrook Terrace, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Luke's Hospital, Kansas City, Missouri
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - PeaceHealth Sacred Heart Medical Center, Springfield, Oregon
  - York Hospital, York, Pennsylvania
  - Dallas VA Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Park CS, Kim HY, Park HJ, Ihm SH, Kim DB, Lee JM, Kim PJ, Park CS, Moon KW, Yoo KD, Jeon DS, Chung WS, Seung KB, Kim JH. Clinical, electrocardiographic, and procedural characteristics of patients with coronary chronic total occlusions. Korean Circ J. 2009 Mar;39(3):111-5. doi: 10.4070/kcj.2009.39.3.111. Epub 2009 Mar 25. PMID 19949597
- [Background] Oesterle SN, Bittl JA, Leon MB, Hamburger J, Tcheng JE, Litvack F, Margolis J, Gilmore P, Madsen R, Holmes D, Moses J, Cohen H, King S 3rd, Brinker J, Hale T, Geraci DJ, Kerker WJ, Popma J. Laser wire for crossing chronic total occlusions: "learning phase" results from the U.S. TOTAL trial. Total Occlusion Trial With Angioplasty by Using a Laser Wire. Cathet Cardiovasc Diagn. 1998 Jun;44(2):235-43. doi: 10.1002/(sici)1097-0304(199806)44:23.0.co;2-k. PMID 9637452
- [Result] Kahn JK. Angiographic suitability for catheter revascularization of total coronary occlusions in patients from a community hospital setting. Am Heart J. 1993 Sep;126(3 Pt 1):561-4. doi: 10.1016/0002-8703(93)90404-w. PMID 8362709
- [Result] Christofferson RD, Lehmann KG, Martin GV, Every N, Caldwell JH, Kapadia SR. Effect of chronic total coronary occlusion on treatment strategy. Am J Cardiol. 2005 May 1;95(9):1088-91. doi: 10.1016/j.amjcard.2004.12.065. PMID 15842978
- [Result] Sirnes PA, Golf S, Myreng Y, Molstad P, Emanuelsson H, Albertsson P, Brekke M, Mangschau A, Endresen K, Kjekshus J. Stenting in Chronic Coronary Occlusion (SICCO): a randomized, controlled trial of adding stent implantation after successful angioplasty. J Am Coll Cardiol. 1996 Nov 15;28(6):1444-51. doi: 10.1016/s0735-1097(96)00349-x. PMID 8917256
- [Result] Moussa I, Di Mario C, Moses J, Reimers B, Di Francesco L, Blengino S, Colombo A. Comparison of angiographic and clinical outcomes of coronary stenting of chronic total occlusions versus subtotal occlusions. Am J Cardiol. 1998 Jan 1;81(1):1-6. doi: 10.1016/s0002-9149(97)00859-x. PMID 9462596
- [Result] Sirnes PA, Golf S, Myreng Y, Molstad P, Albertsson P, Mangschau A, Endresen K, Kjekshus J. Sustained benefit of stenting chronic coronary occlusion: long-term clinical follow-up of the Stenting in Chronic Coronary Occlusion (SICCO) study. J Am Coll Cardiol. 1998 Aug;32(2):305-10. doi: 10.1016/s0735-1097(98)00247-2. PMID 9708454
- [Result] Surmely JF, Tsuchikane E, Katoh O, Nishida Y, Nakayama M, Nakamura S, Oida A, Hattori E, Suzuki T. New concept for CTO recanalization using controlled antegrade and retrograde subintimal tracking: the CART technique. J Invasive Cardiol. 2006 Jul;18(7):334-8. PMID 16816442
- [Result] Suero JA, Marso SP, Jones PG, Laster SB, Huber KC, Giorgi LV, Johnson WL, Rutherford BD. Procedural outcomes and long-term survival among patients undergoing percutaneous coronary intervention of a chronic total occlusion in native coronary arteries: a 20-year experience. J Am Coll Cardiol. 2001 Aug;38(2):409-14. doi: 10.1016/s0735-1097(01)01349-3. PMID 11499731
- [Result] Olivari Z, Rubartelli P, Piscione F, Ettori F, Fontanelli A, Salemme L, Giachero C, Di Mario C, Gabrielli G, Spedicato L, Bedogni F; TOAST-GISE Investigators. Immediate results and one-year clinical outcome after percutaneous coronary interventions in chronic total occlusions: data from a multicenter, prospective, observational study (TOAST-GISE). J Am Coll Cardiol. 2003 May 21;41(10):1672-8. doi: 10.1016/s0735-1097(03)00312-7. PMID 12767645
- [Result] Prasad A, Rihal CS, Lennon RJ, Wiste HJ, Singh M, Holmes DR Jr. Trends in outcomes after percutaneous coronary intervention for chronic total occlusions: a 25-year experience from the Mayo Clinic. J Am Coll Cardiol. 2007 Apr 17;49(15):1611-1618. doi: 10.1016/j.jacc.2006.12.040. Epub 2007 Apr 2. PMID 17433951
- [Result] Valenti R, Migliorini A, Signorini U, Vergara R, Parodi G, Carrabba N, Cerisano G, Antoniucci D. Impact of complete revascularization with percutaneous coronary intervention on survival in patients with at least one chronic total occlusion. Eur Heart J. 2008 Oct;29(19):2336-42. doi: 10.1093/eurheartj/ehn357. Epub 2008 Aug 5. PMID 18682446

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Crossing of Coronary Artery CTO
Started | 163
Completed | 158
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Arm/Group | Crossing of Coronary Artery CTO
Number analyzed (Participants) | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 9
  White | 142
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Procedure Success
Description: Angiographic visualization of any guidewire in a position either distal or proximal to the occlusion depending on the route of access and the absence of in-hospital MACE.
Time Frame: Through hospital discharge, typically 24 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Crossing of Coronary Artery CTO
Number analyzed (Participants) | 163
Participants | 119

2. Secondary Outcome: Frequency of Successful Recanalization
Description: Angiographic confirmation of crossing the chronic total occlusion and restoring blood flow to the affected area.
Time Frame: During Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Crossing of Coronary Artery CTO
Number analyzed (Participants) | 163
Participants | 145

3. Secondary Outcome: Frequency of In-hospital MACE
Description: Any serious adverse experience that includes cardiac death; target lesion revascularization; or post-procedural MI.
Time Frame: Up to hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Crossing of Coronary Artery CTO
Number analyzed (Participants) | 163
Participants | 31

4. Secondary Outcome: Frequency of Perforation
Description: Frequency of perforation during the procedure.
Time Frame: During Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Crossing of Coronary Artery CTO
Number analyzed (Participants) | 163
Participants | 21

5. Secondary Outcome: Frequency of Dissection
Description: Frequency of dissection reported during the procedure
Time Frame: During procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Crossing of Coronary Artery CTO
Number analyzed (Participants) | 163
Participants | 7

6. Secondary Outcome: Mean Procedural Time
Description: The length of the procedure (The first successful insertion of the guide catheter at an arteriotomy site is considered the start of the procedure. A procedure is considered complete once the guide catheter is removed from the arteriotomy site.)
Time Frame: During Procedure
Population: Data collected for 162 of 163 subjects
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Crossing of Coronary Artery CTO
Number analyzed (Participants) | 162
minutes | 118.5 (68.4)

7. Secondary Outcome: Mean Contrast Volume
Description: Volume of contrast administered during procedure
Time Frame: During Procedure
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Crossing of Coronary Artery CTO
Number analyzed (Participants) | 163
milliliters | 287.3 (141.7)

8. Secondary Outcome: Mean Absorbed Radiation Dose in mGy
Description: Absorbed radiation dose in mGy during procedure
Time Frame: During Procedure
Population: Data recorded for 161 of 163 subjects
Measure: Mean (Standard Deviation); unit: milligray (mGy)
Arm/Group | Crossing of Coronary Artery CTO
Number analyzed (Participants) | 161
milligray (mGy) | 2612.7 (1881.3)

9. Secondary Outcome: Procedural Success (Evaluated According to Crossing Technique)
Description: The percentage of subjects with procedure success according to crossing technique
Time Frame: Through hospital discharge
Measure: Count of Participants; unit: Participants
Groups:
- Antegrade Only: Subjects where only an antegrade crossing techinique was used.
- Retrograde Only: Subjects where only a retrograde crossing technique was used
- Antegrade and Retrograde: Subjects were both antegrade and retrograde techniques were used
Arm/Group | Antegrade Only | Retrograde Only | Antegrade and Retrograde
Number analyzed (Participants) | 74 | 9 | 80
Participants | 67 | 6 | 46

ADVERSE EVENTS:
Groups:
- Crossing of Coronary Artery CTO: This is a single arm intent to treat study. A subject is considered enrolled when the subject has given informed consent and meets all inclusion and exclusion criteria, including angiographic inclusion and exclusion criteria, which includes an attempt to cross the target lesion with an investigational device (ASAHI PTCA Guidewire or ASAHI Corsair Microcatheter). Clinical evaluation up to hospital discharge is conducted on all enrolled subjects. The purpose of the clinical follow-up is to determine if the subject has experienced or is experiencing any adverse events.
  Crossing of Coronary Artery CTO: Standard angiographic procedures will be followed for this study. The primary objective of this trial is to evaluate confirmation of placement of any guidewire beyond the chronic total occlusion (CTO) in the true vessel lumen in patients in which at least one Asahi series of guidewires and/or Corsair microcatheter were used.
Arm/Group | Crossing of Coronary Artery CTO
Serious Adverse Events (participants affected / at risk) | 37/163
Other Adverse Events (participants affected / at risk) | 34/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crossing of Coronary Artery CTO (N=163)
Angina pectoris (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 2 (2)
Coronary artery perforation (Cardiac disorders) | 19 (19)
Myocardial infarction (Cardiac disorders) | 5 (5)
Pericardial effusion (Cardiac disorders) | 10 (10)
Pericarditis (Cardiac disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Retroperitoneal haemorrhage (Blood and lymphatic system disorders) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 4 (4)
Multi-organ failure (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Post procedural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 6 (6)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crossing of Coronary Artery CTO (N=163)
Myocardial infarction (Cardiac disorders) | 22 (22)
Catheter site haematoma (General disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish the results of its data 1 year after completion of the Study. Sponsor can review results prior to public release and embargo communications regarding results for a period ≤60 days from the time submitted to the sponsor for review. Sponsor may request in writing (a) deletion of any Confidential Information, (b) reasonable changes requested by Sponsor, or (c) delay of proposed submission for another period ≤90 days in order to protect the potential patentability of any technology.